CLINICAL TRIAL: NCT01667913
Title: The Relative and Absolute Reliability of 6-Minutes Walking Test in Hip Fracture Patients
Brief Title: Reliability of 6-Minutes Walking Test in Hip Fracture Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low inclusion rate we terminated this study with n=20 participants instead of n=50.
Sponsor: Lolland Community, Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Mr. Jan Overgaard, Bachelor in Physiotherapy, Lolland Community, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Hip Fracture study 7/7-12
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Hip Fracture
Keywords: Hip Fracture; 6-minutes walking test; Reliability
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6 minutes walking test (No Intervention)
  Interventions: Other: 6 minutes walking test

INTERVENTIONS:
Other: 6 minutes walking test

SUMMARY:
The purpose of this study is to examine the relative (ICC) and absolute intertester reliability of the 6-Minutes Walking Test in hip fracture patients (N=50) in an outpatient facility. The data collection is conducted by two physiotherapists, who are blinded to each other. The physiotherapists are randomized so they each are doing an equal number of baseline tests.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or above
* Hip fracture patients with a Intra - or Extra Capsular hip fracture
* Testing within 3 - 5 weeks postsurgery in an outpatient facility
* No weightbearing restrictions on the fractured limb
* Normal cognitive level (Mini Mental State Examination(MMSE) - score ≥20 points)
* Participants should not experiencing hip related pain more or less than moderate according to Verbal Ranking Scale when resting
* To have the ability to write and understand danish language

Exclusion Criteria:

- MMSE score ≤19 points

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The 6-Minutes Walking Test | 3 to 5 weeks post surgery
  The 6-Minutes Walking Test performed according to International Guidelines, will be performed on hip fracture patients 3 to 5 weeks after surgery. The testing will be conducted on the same person by two physiotherapists with a one day pause in between test sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Overgaard, Bachelor, Principal Investigator — Sector of Health and Older, Department of Rehabilitation, Lolland Community, Denmark; Morten T Kristensen, Ph.d, Study Director — Department of Physical Therapy and Orthopedic Surgery, Copenhagen University Hospital at Hvidovre, Denmark
Locations (1):
- Health Center Maribo, Maribo, Denmark

REFERENCES:
- See also: Protocol for the 6-Minutes Walking Test — http://www.thoracic.org/statements/resources/pfet/sixminute.pdf